CLINICAL TRIAL: NCT00777270
Title: Continuous Versus Interrupted Sutures for Repair of Episiotomy or Second Degree Tears: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Principe de Asturias (Other)
Responsible Party: Pedro Valenzuela, Fundación Hospital Principe de Asturias
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIS-PI051023
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2008-10-22 (Estimated); Status verified 2008-10

CONDITIONS: Pain
Keywords: episiotomy; perineal lesion; vaginal trauma
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 continuous (Experimental): continuous suture technique with continuous non-locking suture in the vagina, perineum and subcutaneous tissue.
  Interventions: Procedure: repair of episiotomy or second degree tears
- 2 interrupted (Experimental): interrupted technique with continuous locking suture of the vagina, interrupted sutures in the perineum muscle and interrupted transcutaneous suture
  Interventions: Procedure: repair of episiotomy or second degree tears

INTERVENTIONS:
Procedure: repair of episiotomy or second degree tears — continuous suture technique with continuous non-locking suture in the vagina, perineum and subcutaneous tissue.
  Other Names: (Vicryl Rapid; Ethicon)
  Arms: 1 continuous
Procedure: repair of episiotomy or second degree tears — interrupted technique with continuous locking suture of the vagina, interrupted sutures in the perineum muscle and interrupted transcutaneous suture
  Other Names: (Vicryl Rapid; Ethicon).

SUMMARY:
The best technique for this repair would be that which requires least time in realisation, least consumption of material for the repair and that which produces less pain at short and long-term permitting the resumption of intercourse quicker and with less pain thereby requiring less necessity to take out the stitches and less frequency of re stitching. The investigators research is looking for a technique for repairing the perineum more advantageously.

DETAILED DESCRIPTION:
445 women who participated in the project had undergone normal deliveries with episiotomy or second-grade tearing of the perineum. One group was repaired with continuous non-locking suture in the vagina, perineum and subcutaneous tissue. The other group used continuous locking suture of the vagina, interrupted sutures in the perineum muscle and interrupted transcutaneous suture. The threads used for stitching were identical in both groups. The same questions were asked concerning the sensation of pain and the use of painkillers, the second and the tenth day and at the three months.

ELIGIBILITY:
Inclusion Criteria:

* vaginal childbirth
* at least 37 weeks of gestation
* assistance by one of the 4 matrons who participated in the project
* have been subjected to an episiotomy or the appearance of tearing that affected skin and muscle
* The newborn child had to be alive, viable

Exclusion Criteria:

* instrumentation
* produce injury in the anal sphincter or in the rectum.
* serious congenital malformations.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pain at that moment ("pain now") | the second and the tenth day and at the three months.

SECONDARY OUTCOMES:
If sexual intercourse had been re initiated, how long after childbirth, if pain had been experienced the first time and if this continued. | at the three months.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Valenzuela, MD, Principal Investigator — Hospital Prínicpe de Asturias
Locations (1):
- Fundación Hospital Príncipe de Asturias, Alcalá de Henares, Madrid, Spain

REFERENCES:
- [Result] Kettle C, Hills RK, Jones P, Darby L, Gray R, Johanson R. Continuous versus interrupted perineal repair with standard or rapidly absorbed sutures after spontaneous vaginal birth: a randomised controlled trial. Lancet. 2002 Jun 29;359(9325):2217-23. doi: 10.1016/S0140-6736(02)09312-1. PMID 12103284
- [Result] Fleming N. Can the suturing method make a difference in postpartum perineal pain? J Nurse Midwifery. 1990 Jan-Feb;35(1):19-25. doi: 10.1016/0091-2182(90)90053-8. PMID 2406391